CLINICAL TRIAL: NCT00445484
Title: Revlimid to Augment Efficacy of Prevnar Vaccines in Patients With Relapsed or Refractory Myeloma
Brief Title: Lenalidomide and Vaccine Therapy in Treating Patients With Relapsed or Refractory Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: J06102 CDR0000532944; P30CA006973 (NIH); JHOC-J06102; JHOC-NA_00006008; CELGENE-CC-5013
Record Dates: First submitted 2007-03-07; First posted 2007-03-09 (Estimated); Results first posted 2015-07-24 (Estimated); Last update posted 2015-08-24 (Estimated); Status verified 2015-08

CONDITIONS: Multiple Myeloma and Plasma Cell Neoplasm
Keywords: stage II multiple myeloma; stage III multiple myeloma; refractory multiple myeloma
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — Pneumococcal Vaccines; Lenalidomide

ARMS (2):
- Group 1 (Experimental): Patients receive oral lenalidomide on days 1-21. Treatment repeats every 28 days for up to 7 courses in the absence of disease progression or unacceptable toxicity. Patients receive pneumococcal polyvalent vaccine intramuscularly (IM) 14 days prior to beginning lenalidomide and again in approximately 2 months (after the first dose of the vaccine).
  Interventions: Biological: pneumococcal polyvalent vaccine; Drug: lenalidomide
- Group 2 (Experimental): Patients receive lenalidomide as in group 1. Patients receive pneumococcal polyvalent vaccine IM approximately 45 days after beginning lenalidomide and again in approximately 2 months (after the first dose of the vaccine).
  Interventions: Biological: pneumococcal polyvalent vaccine; Drug: lenalidomide

INTERVENTIONS:
Biological: pneumococcal polyvalent vaccine — Given intramuscularly
Drug: lenalidomide — Given orally

SUMMARY:
RATIONALE: Biological therapies, such as lenalidomide, may stimulate the immune system in different ways and stop cancer cells from growing. Vaccines may help the body build an effective immune response to kill cancer cells. Giving lenalidomide together with vaccine therapy may make a stronger immune response and kill more cancer cells.

PURPOSE: This phase II trial is studying how well giving lenalidomide together with vaccine therapy works in treating patients with relapsed or refractory multiple myeloma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine whether lenalidomide can augment the efficacy of pneumococcal polyvalent vaccine as it correlates with lenalidomide-induced antitumor efficacy in patients with relapsed or refractory multiple myeloma.

Secondary

* Determine the antibody responses to pneumococcal serotypes in patients treated with this regimen.
* Determine T-cell responses to the carrier protein CRM 197 in patients treated with this regimen.
* Determine the ability of lenalidomide to augment in vivo immune responsiveness as measured by cutaneous delayed-type hypersensitivity (DTH) reactions to Candida and tetanus in these patients.
* Determine the ability of lenalidomide to prime and/or boost systemic vaccine responses in both peripheral blood lymphocytes and marrow lymphocytes in these patients.

OUTLINE: Patients are assigned to 1 of 2 treatment groups.

* Group 1: Patients receive oral lenalidomide on days 1-21. Treatment repeats every 28 days for up to 7 courses in the absence of disease progression or unacceptable toxicity. Patients receive pneumococcal polyvalent vaccine intramuscularly (IM) 14 days prior to beginning lenalidomide and again in approximately 2 months (after the first dose of the vaccine).
* Group 2: Patients receive lenalidomide as in group 1. Patients receive pneumococcal polyvalent vaccine IM approximately 45 days after beginning lenalidomide and again in approximately 2 months (after the first dose of the vaccine).

After completion of study treatment, patients are followed at 30 days.

PROJECTED ACCRUAL: A total of 40 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of multiple myeloma (MM) meeting all of the following criteria:

  * Relapsed or refractory disease
  * Previously received ≥ 2 courses of antimyeloma treatment
* Measurable levels of myeloma paraprotein in serum (> 0.5 g/dL) or urine (> 0.2 g/24-hour urine collection) OR serum-free light-chain disease

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Absolute neutrophil count ≥ 1,000/mm^3
* Platelet count ≥ 75,000/mm^3
* Creatinine ≤ 2.5 mg/dL
* Bilirubin ≤ 2.0 mg/dL
* AST and ALT ≤ 3 times upper limit of normal
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use 2 methods of highly effective contraception ≥ 4 weeks before, during, and for 4 weeks after completion of study therapy
* No other malignancy within the past 5 years except treated basal cell or squamous cell carcinoma of the skin or carcinoma in situ of the cervix or breast
* No serious medical condition, laboratory abnormality, or psychiatric illness that would preclude study treatment or put patient at unacceptable risk
* No known hypersensitivity to thalidomide or lenalidomide

  * No development of erythema nodosum in the presence of a reaction characterized by a desquamating rash while taking thalidomide or similar drugs
* No known hypersensitivity to any component of the pneumococcal polyvalent vaccine, including diphtheria toxin or CRM 197
* No known HIV positivity
* No infectious hepatitis type A, B, or C

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No more than 3 prior treatment regimens for MM
* More than 6 months since prior lenalidomide
* More than 28 days since prior experimental drug or therapy
* More than 1 month since prior systemic antimyeloma therapy
* More than 1 month since prior and no concurrent systemic corticosteroids
* No other concurrent anticancer agents or treatments or investigational agents
* No concurrent thalidomide
* No concurrent radiotherapy
* No other concurrent immune therapy or immunomodulatory agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2007-01; Primary Completion 2009-04 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ivan Borrello, MD, Study Chair — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States

REFERENCES:
- [Result] Noonan K, Rudraraju L, Ferguson A, Emerling A, Pasetti MF, Huff CA, Borrello I. Lenalidomide-induced immunomodulation in multiple myeloma: impact on vaccines and antitumor responses. Clin Cancer Res. 2012 Mar 1;18(5):1426-34. doi: 10.1158/1078-0432.CCR-11-1221. Epub 2012 Jan 12. PMID 22241792

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group 2 | Group 1
Started | 11 | 11
Completed | 7 | 10
Not Completed | 4 | 1

BASELINE CHARACTERISTICS:
Population: A total of 22 patients were enrolled, 11 in each cohort. Patients who showed evidence of disease progression while on study were not included in subsequent analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2 | Total
Number analyzed (Participants) | 11 | 11 | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.3 (9.0) | 65.8 (10.3) | 66.0 (9.5)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 6 | 11
  >=65 years | 6 | 5 | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 4 | 11
  Male | 4 | 7 | 11
Region of Enrollment [Number; unit: participants]
  United States | 11 | 11 | 22

OUTCOME MEASURES:

1. Primary Outcome: 6B Antibody Response to Prevnar Vaccine in Peripheral Blood
Description: Serum IgG levels against the PVC serotype were measured by ELISA
Time Frame: basline and 8 weeks after second vaccination
Population: Patients who showed evidence of disease progression while on study were not included in the analysis.
Measure: Mean (Standard Error); unit: fold change
Groups:
- Vaccine Started 14 Days Prior to Lenalidomide: Patients receive oral lenalidomide on days 1-21. Treatment repeats every 28 days for up to 7 courses in the absence of disease progression or unacceptable toxicity. Patients receive pneumococcal polyvalent vaccine intramuscularly (IM) 14 days prior to beginning lenalidomide and again in approximately 2 months (after the first dose of the vaccine).
  pneumococcal polyvalent vaccine: Given intramuscularly
  lenalidomide: Given orally
- Vaccine Started 45 Days After Lenalidomide: Patients receive lenalidomide as in group 1. Patients receive pneumococcal polyvalent vaccine IM approximately 45 days after beginning lenalidomide and again in approximately 2 months (after the first dose of the vaccine).
  pneumococcal polyvalent vaccine: Given intramuscularly
  lenalidomide: Given orally
Arm/Group | Vaccine Started 14 Days Prior to Lenalidomide | Vaccine Started 45 Days After Lenalidomide
Number analyzed (Participants) | 8 | 5
fold change | 3.69 (1.1) | 7.58 (3.0)

2. Primary Outcome: 14F Antibody Response to Prevnar Vaccine in Peripheral Blood
Description: Serum IgG levels against the PVC serotype were measured by ELISA
Time Frame: basline and 8 weeks after second vaccination
Population: Patients who showed evidence of disease progression while on study were not included in the analysis.
Measure: Mean (Standard Error); unit: fold change
Arm/Group | Vaccine Started 14 Days Prior to Lenalidomide | Vaccine Started 45 Days After Lenalidomide
Number analyzed (Participants) | 5 | 8
fold change | 9.42 (5.0) | 11.95 (3.8)

3. Primary Outcome: 19F Antibody Response to Prevnar Vaccine in Peripheral Blood
Description: Serum IgG levels against the PVC serotype were measured by ELISA
Time Frame: basline and 8 weeks after second vaccination
Population: Patients who showed evidence of disease progression while on study were not included in the analysis.
Measure: Mean (Standard Error); unit: fold change
Arm/Group | Vaccine Started 14 Days Prior to Lenalidomide | Vaccine Started 45 Days After Lenalidomide
Number analyzed (Participants) | 8 | 5
fold change | 2.025 (0.64) | 2.12 (0.4)

4. Primary Outcome: 23F Antibody Response to Prevnar Vaccine in Peripheral Blood
Description: Serum IgG levels against the PVC serotype were measured by ELISA
Time Frame: basline and 8 weeks after second vaccination
Population: Patients who showed evidence of disease progression while on study were not included in the analysis.
Measure: Mean (Standard Error); unit: fold change
Arm/Group | Vaccine Started 14 Days Prior to Lenalidomide | Vaccine Started 45 Days After Lenalidomide
Number analyzed (Participants) | 8 | 5
fold change | 4.1 (1.8) | 2.42 (1)

ADVERSE EVENTS:
Arm/Group | Group 1 | Group 2
Serious Adverse Events (participants affected / at risk) | 1/11 | 0/11
Other Adverse Events (participants affected / at risk) | 1/11 | 1/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (N=11) | Group 2 (N=11)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (N=11) | Group 2 (N=11)
Lower back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Shortness of breath on exertion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Renal insufficiency (Renal and urinary disorders) | 0 (0) | 1 (1)
Hypertension (Cardiac disorders) | 0 (0) | 1 (1)
Hyperlipidemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes